CLINICAL TRIAL: NCT05677243
Title: Observational Study on the Treatment of Trigeminal Neuralgia by Radiosurgery
Acronym: NATURE
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Princesse Grace (Other)
Collaborators: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 21-19
Record Dates: First submitted 2022-12-15; First posted 2023-01-10 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Trigeminal Neuralgia
Keywords: Trigeminal Neuralgia; Radiosurgery; LINAC; Pain relief; Hypesthesia
MeSH Terms: conditions — Trigeminal Neuralgia; Hypesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study aims to evaluate the outcome of patient treated by radiosurgery on LINAC with high dose rate for classical trigeminal neuralgia

DETAILED DESCRIPTION:
This retrospective and prospective case-series hospital-based study will be conducted in all patients with trigeminal neuralgia treated by radiosurgery on LINAC at the Centre Hospitalier Princesse Grace from april 2018 to january 2028. Patients will be treated with frameless technic and receive 90 Gy delivered with high dose rate on the intra cisternal portion of the trigeminal nerve.

ELIGIBILITY:
Inclusion Criteria:

* Classical trigeminal neuralgia according the International Classification of Headache Disorders
* Trigeminal neuralgia resistant to the maximum tolerated medical therapy, with pain intensity according to the Barrow Neurological Institute (BNI) score IV or V.
* Patients aged > 18

Exclusion Criteria:

* Patients suffering from secondary Trigeminal neuralgia (tumour in the cerebellopontine angle, arteriovenous malformation or multiple sclerosis)
* Previous history of radiosurgery procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients with trigeminal neuralgia treated by radiosurgery on LINAC
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2036-12 (Estimated)

PRIMARY OUTCOMES:
Pain relief | 24 months
  Barrow Neurological Institute pain intensity scale - score I to V - V is the worst
  Barrow Neurological Institute (BNI) pain intensity scale
  Barrow Neurological Institute (BNI) pain intensity scale

SECONDARY OUTCOMES:
Toxicity of radiosurgery | 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10 years
  Common Terminology Criteria for Adverse Events version 5.0 - grade 1 to 5 - 5 is the worst
Variation of quality of life | 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10 years
  Short Form 36 Health Survey - score 0 to 100 - 0 is the worst

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Princesse Grace, Monaco, Monaco